CLINICAL TRIAL: NCT02993653
Title: Definitive Treatment Protocol for High-dose Intensity-modulated Radiotherapy (IMRT) With Intracavitary Radiotherapy in Locally Advanced Cervical Cancer: A Phase II Trial
Brief Title: Intensity-modulated Radiotherapy Protocol in Cervix Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Jong Hoon Lee, Professor, Seoul St. Mary's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VINPI1501
Record Dates: First submitted 2016-12-11; First posted 2016-12-15 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Radiation
MeSH Terms: interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intensity-modulated radiotheapy arm (Experimental): Intensity-modulated radiotheapy with stereotactic boost or intracavitary radiotherapy
  Interventions: Radiation: High-dose Intensity-modulated radiotherapy

INTERVENTIONS:
Radiation: High-dose Intensity-modulated radiotherapy — Pelvic High-dose Intensity-modulated radiotherapy with stereotactic radiotherapy or intracavitary radiotherapy

SUMMARY:
Definitive treatment protocol for high-dose intensity-modulated radiotherapy (IMRT) with intracavitary radiotherapy in locally advanced cervical cancer: A phase II trial

DETAILED DESCRIPTION:
Radiotherapy

1. intensity-modulated radiotherapy of whole pelvis: 60 Gy in 30 fx Re-simulation with pelvic Magnetic resonance imaging at 46 Gy in 23 fx and intensity-modulated radiotherapy on the gross cervical and nodal tumor (initially Positron emission tomography-positive), 14 Gy in 7 fx
2. intensity-modulated radiotherapy boost of gross cervical tumor or Intra-cavitary radiotherapy (ICR)

   * Re-staging pelvic Magnetic resonance imaging , if complete response occurs Intra-cavitary radiotherapy to A point, 25 Gy in 5 fx for 2 weeks
   * Re-staging pelvic Magnetic resonance imaging I, partial response or stable disease occurs intensity-modulated radiotherapy boost , 10 Gy in 4 fx to the gross cervical tumor for 1 week

ELIGIBILITY:
Inclusion Criteria:

1. FIGO II-IVA Patients with untreated and histologically confirmed carcinoma of the uterine cervix
2. Patients with Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1
3. Patients with adequate bone marrow function: Absolute nutrophil count (ANC) greater than or equal to 1,500/mcl, platelets greater than or equal to 100,000/mcl at the beginning
4. Patients with adequate renal function: creatinine equal to or less than 2.0 mg/mL
5. Patients who have signed an approved informed consent and authorization

Exclusion Criteria:

1. Patients with recurrent cervical cancer
2. Patients who have diagnosis of other malignance tumors except papillary or follicular thyroid cancer or skin cancer
3. Patients with metastatic lymphadenopathies other than pelvis (e.g. inguinal, paraaortic, supraclavicular, or mediastinal node)
4. Patients with distant organ metastasis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 30 months
  Progression means locoregional recurrence, distant metastasis, and local tumor pregression

SECONDARY OUTCOMES:
Overall survival | 30 months
Treatment-related adverse events are assessed by CTCAE v4.0. | acute within 3 months and chronic after 3 months after radiotherapy
  Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Jong Hoon Lee, MD, Principal Investigator — St. Vincent's Hospital, South Korea
Locations (1):
- Lee Jong Hoon, Suwon, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kang HB, Kim SH, Lee JH, Lee HC, Kang NK, Lee JH. MRI-based volumetric tumor parameters before and during chemoradiation predict tumor recurrence and patient survival in locally advanced cervical cancer: a subgroup analysis of a phase II prospective trial. Int J Clin Oncol. 2024 May;29(5):620-628. doi: 10.1007/s10147-024-02490-7. Epub 2024 Mar 26. PMID 38530569
- [Derived] Lee HC, Jeong JW, Lee JH, Kim SH, Park DC, Yoon JH, Kim SI, Lee JH. High-dose (60 Gy) intensity-modulated radiotherapy with concurrent weekly cisplatin followed by intracavitary radiation in locally advanced cervical cancer: A phase II prospective clinical trial. Gynecol Oncol. 2023 Oct;177:142-149. doi: 10.1016/j.ygyno.2023.08.018. Epub 2023 Sep 7. PMID 37689018